CLINICAL TRIAL: NCT05837260
Title: A Multicentre Prospective Study Investigating the Utility of ctDNA as a Biomarker of Disease Burden, Genetic Heterogeneity and Tumour Evolution in Advanced Thyroid Cancer
Brief Title: Investigating Utility of ctDNA and Tumour Evolution in Advanced Thyroid Cancer
Acronym: NOMINATE
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5637
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Patients with newly diagnosed iodine refractory thyroid cancer on surveillance
  Interventions: Other: Sample collection only
- Cohort 2: Patients with locally advanced and / or metastatic (Stage 3 & 4) medullary thyroid cancer
  Interventions: Other: Sample collection only
- Cohort 3: Patients with iodine refractory thyroid cancer or advanced/metastatic unresectable MTC due to commence systemic treatment or already on systemic treatment
  Interventions: Other: Sample collection only
- Cohort 4: Patients with newly diagnosed anaplastic thyroid cancer
  Interventions: Other: Sample collection only

INTERVENTIONS:
Other: Sample collection only — Sample collection only

SUMMARY:
Although most thyroid cancers are treated and cured successfully there are still 30% who recur after many years. This will eventually progress and at this point may become incurable with treatment options including complex and high risk surgery. The overall efficacy of systemic treatment in advanced thyroid cancer has a good initial response in most patients but not all. The study will collect tissues and blood samples for various protein analysis, nucleic acid extraction and live cell analysis in order to try and detect the presence of plasma ctDNA at baseline of eligible patients.

DETAILED DESCRIPTION:
The treatment decisions are based on relying on radiological parameters such as using the RECIST criteria and measuring the rise in certain serum tumour biomarkers. However, the disadvantage of this is that this method can take many months to detect a change in disease volume. An improved understanding of genetics and cancer and potential gene sequencing can help achieve personalised treatment for patients. However, there are many questions and issues that still need to be answered and require urgent attention before being able to achieve optimate patient stratification. We need to identify better tumour biomarkers to detect disease progression, show real time response to treatment and understand why tumours evolve to becoming more aggressive. This study hopes to address these issues by proposing a multicentre prospective study to investigate the presence and role of ctDNA in advanced thyroid cancer including differentiated thyroid cancer , medullary thyroid cancer and Anaplastic Thyroid Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older. (all cohorts)
* Patients diagnosed with radioiodine refractory differentiated thyroid carcinoma (RR-DTC) under surveillance. (cohort 1)
* Patients with newly diagnosed resectable locally advanced medullary thyroid cancer Or Patients with newly diagnosed metastatic medullary thyroid cancer for surveillance Or Patients with locally advanced or metastatic medullary thyroid cancer on surveillance (cohort 2)
* Patients with RR-DTC starting systemic therapy Or Patients with RR-DTC on systemic therapy Or Patients with MTC starting systemic therapy Or Patients with MTC on systemic therapy (cohort 3)
* Patients with newly diagnosed anaplastic thyroid cancer (cohort 4)
* Availability of tissue from one archival diagnostic tumour tissue block or be willing to have biopsy of accessible disease (all cohorts)
* Patients must be willing to undergo standard monitoring and treatment as recommended by their clinical team (all cohorts)
* Ability to give informed consent for biological sample collection. (all cohorts)

Exclusion Criteria:

* Previous or concurrent illness, which in the investigator's opinion would interfere with collection of the complete sample collection
* Any invasive malignancy within previous 5 years (other than non-melanomatous skin carcinoma or carcinoma in situ)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-02-07 (Estimated); Study Completion 2027-02-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the proposed study is to determine the sensitivity of detecting the presence of plasma ctDNA in patients with advanced and recurrent thyroid cancer | 5 years
  The primary objective of the proposed study is to determine the sensitivity of detecting the presence of plasma ctDNA in patients with advanced and recurrent thyroid cancer

SECONDARY OUTCOMES:
Specificity of the absence of plasma ctDNA in patients with advanced and recurrent thyroid cancer at baseline | 5 years
  Specificity of the absence of plasma ctDNA in patients with advanced and recurrent thyroid cancer at baseline
Association of ctDNA levels as biomarker of disease burden compared with standard biochemical markers and radiological response | 5 years
  Association of ctDNA levels as biomarker of disease burden compared with standard biochemical markers and radiological response
Changes in ctDNA levels as biomarker of disease burden compared with standard biochemical markers and radiological response | 5 years
  Changes in ctDNA levels as biomarker of disease burden compared with standard biochemical markers and radiological response
ctDNA as a biomarker of response to systemic therapy (levels and timing) compared with standard biochemical markers and radiological response in patients starting/during systemic therapy | 5 years
  ctDNA as a biomarker of response to systemic therapy (levels and timing) compared with standard biochemical markers and radiological response in patients starting/during systemic therapy
ctDNA as a biomarker of progression free and overall survival | 5 years
  ctDNA as a biomarker of progression free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kate Newbold, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided